CLINICAL TRIAL: NCT02106130
Title: A Randomized, Open-label, Multiple Dose, Two-treatment, Two-period, Two-sequence Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Mosapride Citrate and Rebamipide After Oral Administration in Healthy Volunteers
Brief Title: A Drug Interaction Study of Mosapride and Rebamipide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID_MotiReb_1201
Record Dates: First submitted 2014-03-12; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Mosapride citrate; Rebamipide; pharmacokinetic drug drug interaction; oral administration; healthy male subjects
MeSH Terms: interventions — rebamipide; mosapride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- R - R+M (Experimental): R : Rebamipide 100mg, M : Mosapride citrate 5mg, All drugs will be administered orally.
  Interventions: Drug: Rebamipide; Drug: Mosapride citrate
- R+M - R (Experimental): R : Rebamipide 100mg, M : Mosapride citrate 5mg, All drugs will be administered orally.
  Interventions: Drug: Rebamipide; Drug: Mosapride citrate
- M - R+M (Experimental): R : Rebamipide 100mg, M : Mosapride citrate 5mg, All drugs will be administered orally.
  Interventions: Drug: Rebamipide; Drug: Mosapride citrate
- R+M - M (Experimental): R : Rebamipide 100mg, M : Mosapride citrate 5mg, All drugs will be administered orally.
  Interventions: Drug: Rebamipide; Drug: Mosapride citrate

INTERVENTIONS:
Drug: Rebamipide — oral administration, 3 times/day
  Other Names: Mucosta® Tab.
Drug: Mosapride citrate — oral administration, 3 times/day
  Other Names: Gasmotin® tab.

SUMMARY:
The investigators investigate the potential pharmacokinetic drug-drug interaction between Mosapride citrate 5 mg and Rebamipide 100 mg in healthy male volunteers who receive Mosapride citrate 5 mg, Rebamipide 100 mg, and both together in a 2 period repeatedly.

DETAILED DESCRIPTION:
To evaluate the safety, drug-tolerance, pharmacokinetics of Mosapride citrate 5 mg or Rebamipide 100 mg monotherapy or Mosapride citrate 5 mg and Rebamipide 100 mg combination in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, age 20 to 45 years
2. Body weight ≥ 55kg (male), ≥ 50kg (female)
3. Body weight index (BMI) 18.5 ~ 25
4. Acceptable serum test, hematologic test, blood chemistry examination, urin test and ECG, physical examination during screening
5. Subject decided to participate voluntarily and gave written Informed consent to comply with the instructions after listening to and fully understanding the detailed explanation about this trial.

Exclusion Criteria:

1. Subject has clinically significant liver, kidney, neurologic, immunologic, respiratory, endocrine disease or hematologic·oncologic disease, cardiovascular disease or psychiatric disease (mood disorder, compulsive disorder etc.) or such medical history (including subject with hepatitis virus in case of liver disease).
2. Subject has history of gastrointestinal disease (such as Crohn's disease, ulcer, acute or chronic pancreatitis etc.) or gastrointestinal surgery (except simple appendectomy or hernia operation) that can affect the absorption of the study drug.
3. Subject has hypersensitivity reaction to drug (aspirin, antibiotics, including study durgs, etc.) or history of clinically significant hypersensitivity reaction.
4. Systolic blood pressure > 150mmHg or <90mmHg, Diastolic blood pressure >100mmHg or <50mmHg(Sitting blood pressure) during the screening procedure
5. Subject has history of drug abuse or tested positive to abused drug in the urine drug screening test.
6. For women, pregnant or breastfeeding woman or woman who was confirmed to be pregnant in the pregnancy test
7. Subject takes caffeine-containing food 5 cups per day
8. Subject continually drinks (in excess of 210g/week)
9. Subject smokes 10 cigarettes or more in one day
10. Subject took any prescribed drug or oriental medicine within 2 weeks prior to the first medication or any over-the-counter (OTC) drug within 1 week prior to the first medication (however, the subject can be included if other criteria are met according to the discretion of the investigator).
11. A subject who takes grapefruit, grapefruit juice, or grapefruit-containing products within 30 days prior to the first dosing
12. Subject participated in another study and received medication within 2 months prior to the first medication day.
13. Subject received whole blood transfusion (500 mL) within 2 months prior to the first medication or blood transfusion within 1 month prior to the first medication.
14. Subject was judged not to be eligible according to the discretion of the investigator for other reasons.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of Mosapirde citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Cmax,ss of Mosapirde citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
AUCτ,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Cmax,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose

SECONDARY OUTCOMES:
AUClast,ss of Mosapride citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
AUCinf,ss of Mosapride citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Tmax,ss of Mosapride citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
t1/2 of Mosapride citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Cmin,ss of Mosapride citrate 5mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
AUClast,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
AUCinf,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Tmax,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
t1/2 of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose
Cmin,ss of Rebamipide 100mg | D-1 D2, D7, D9: pre-dose / D3~4, D10~11: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 25 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Chun-ok Kim, MD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea